CLINICAL TRIAL: NCT06651450
Title: Investigation of Perioperative Electrocardiographic Changes in Laparoscopic Cholecystectomy Surgery
Brief Title: Electrocardiographic Changes in Cholecystectomy Surgery
Status: Enrolling by invitation | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Ali Genc, Assistant professor, Tokat Gaziosmanpasa University
Other Study IDs: 24-KAEK-215
Record Dates: First submitted 2024-10-16; First posted 2024-10-21 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-08

CONDITIONS: Laparoscopic Cholecystectomy; Vector Electrocardiography
Keywords: Electrocardiography; general anesthesia; pneumoperitoneum; vectorcardiography; cardiac arrhythmias
MeSH Terms: conditions — Pneumoperitoneum; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent laparoscopic cholecystectomy surgery: Effects of increasing IAB on frontal plane QRS-T angle, QT and QTc in ECG at different stages of surgery

SUMMARY:
Laparoscopic (closed) surgery provides several advantages over open surgery, such as smaller surgical incisions, postoperative recovery, and shorter hospital stay. However, increased intra-abdominal pressure (IAP) during surgery may have adverse effects on some systems such as circulation and respiration. Increased IAP may reduce blood return to the heart. Some studies have shown that some values calculated from surface electrocardiography are associated with changes in heart rhythm. Changes in blood pressure, nervous, and hormonal systems that may be seen due to increased IAP in laparoscopic surgery may cause arrhythmias in patients.Therefore, researchers aimed to investigate the effects of increased IAP on electrocardiography in patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy has been shown to have advantages such as less postoperative pain, early onset of bowel movements, shortening of hospital stay, early return to daily activities and better aesthetic results compared to open surgery. However, increased intra-abdominal pressure (IAP) can negatively affect the respiratory, circulatory, neuroendocrine and central nervous systems. Increased IAP can compress the vena cava and abdominal aorta, causing deterioration in the perfusion of other organs, especially the kidneys and spleen. In addition, this pathological process reduces the preload of the heart, stroke volume, cardiac output and increases central venous pressure, pulmonary capillary wedge pressure, pulmonary artery pressure and left ventricular afterload. IAP can also affect the pressure in the coronary arteries and impair the nutrition of the heart. It should be noted that increased IAP has also been identified as an independent risk factor for mortality in critically ill patients. The QT interval, which represents the time required for ventricular depolarization and repolarization on the ECG, is the time interval from the beginning of the QRS complex to the end of the T wave. Since the Qt interval is affected by the heart rate, it is called QT corrected according to the heart rate, QTc. Prolongation of the peroperative QT and QTc intervals can result in serious complications such as serious arrhythmias, ventricular tachycardia, ventricular fibrillation, and cardiac arrest. Variable QT intervals have been associated with heterogeneous repolarization and ventricular arrhythmias. The frontal plane QRS-T angle is expressed as the absolute difference between the QRS and T wave axes. The frontal plane QRS-T angle, a parameter that can be easily calculated from the 12-lead surface ECG, is considered a marker of ventricular repolarization heterogeneity. Increased ventricular repolarization heterogeneity is associated with an increased risk of arrhythmogenesis. Studies have shown that increased frontal plane QRS-T angle leads to an increased risk of cardiovascular and arrhythmic events and is associated with an increased risk of mortality. Previous publications have reported that the frontal plane QRS-T angle value is stronger, more renewable, and less affected by external factors than the QT/QTc value in showing ventricular repolarization. A wider frontal plane QRS-T angle is considered a strong and independent risk indicator for cardiac morbidity and mortality compared to other traditional cardiovascular risk factors such as the length of the QT interval and electrocardiographic risk indicators. The increase in IAP in laparoscopic surgeries, anesthetic drugs, patient positions, and neuroendocrine response may increase the risk of arrhythmia in the patient. There are many studies on the effects of laparoscopic surgeries, anesthetic drugs, and anesthesia methods that increase IAP on the QT/QTc duration, and there are a limited number of studies in the literature on the effects of another repolarization parameter, the frontal plane QRS-T angle. In this study, researchers investigated perioperative frontal QRS-T angle change and risk of arrhythmia predisposition in patients undergoing laparoscopic cholecystectomy under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 who wish to participate in the study and undergo laparoscopic cholecystectomy

Exclusion Criteria:

* Cardiovascular diseases (coronary artery disease, atrial fibrillation, atrial flutter, heart failure, pacemaker, ICD, CRT, bundle branch block)
* Serious respiratory diseases
* Electrolyte disorders
* Renal failure
* Metabolic diseases
* Advanced psychiatric diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People between the ages of 18-65 who are scheduled to undergo laparoscopic cholecystectomy are included in the study. When calculating the sample size; when the effect size obtained from the previous study was accepted as 0.4, the type 1 error value as 0.05, and the power as 0.80, it was determined that the sample size for the study was sufficient with 44 patients. Considering the losses that may occur during follow-up, it was planned to conduct the study with 48 patients with a 10% increase.
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
frontal plane QRS-T angle, QT and QTc interval | EECG recordings will be taken immediately before surgery, before and immediately after intra-abdominal CO2 insufflation, 2 minutes after reverse Trendelenburg, immediately after the patient is awakened, and at the 2nd hour after surgery.
  The frontal plane QRS-T angle, which is accepted as the ventricular repolarization parameter, describes the angle between the QRS and T axes calculated from the surface ECG.The QT interval, which represents the time required for ventricular depolarization and repolarization on the ECG, is the time interval from the beginning of the QRS complex to the end of the T wave.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Genc A, Ozsoy U, Sahin AT, Gurler Balta M, Kolukcu V, Genc Tapar G, Karaman T, Karaman S. Intra-abdominal hypertension and reverse Trendelenburg position increase frontal QRS-T angle in laparoscopic cholecystectomy: An observational study. Medicine (Baltimore). 2025 Mar 14;104(11):e41934. doi: 10.1097/MD.0000000000041934. PMID 40101078